CLINICAL TRIAL: NCT04600401
Title: Efficacy of Positive Mental Health Program for Adults
Brief Title: Efficacy of Positive Mental Health Program for Adults - Study Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carme Ferré Grau (Other)
Collaborators: Administração Regional de Saúde do Norte, Portugal (Other)
Responsible Party: Sponsor-Investigator, Carme Ferré Grau, Clinical Professor, University Rovira i Virgili
Organization: University Rovira i Virgili (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020PMHP.PT
Record Dates: First submitted 2020-05-15; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Mental Health
Keywords: mental health; program; randomized controlled trial; nursing; health promotion; adult
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either the Mentis Plus+ program (experimental group) or the control group (stand-by group).
Who Masked: Investigator
Masking Description: the researcher, who will collect the outcome assessments and assume data entry and analysis, will stay blinded to treatment allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants integrate the Mentis Plus+ program (Experimental): Mentis Plus+ Program was developed based in The Multifactorial Model of Positive Mental Health and its construction resulted from a systematic literature review and validation through focus group. The duration of the Mentis Plus+ program depends on the number of the six factors to be worked on. The Mentis Plus+ lasts at least 7 weeks (1 session per week, lasting 1 hour) and can work individually or in groups (2-12 people). There will be 2 initial sessions of 1 hour each and 3 sessions for each factor to work with duration of 1 hour. Still, a final session and a follow-up session (3-6 months after the program) will be held.
  Interventions: Other: Mentis Plus+ (Experimental Group)
- Participants on a waiting list (Control Group) (No Intervention): Participants in the control group were told they were on a waiting list for 3-6 months, as a minimum, before they integrate the Mentis Plus+ program. Given the preventive nature of this study, a waiting list control group won't bring risks or damages to participants

INTERVENTIONS:
Other: Mentis Plus+ (Experimental Group) — Each factor can be considered a module, so it is a modular program. So, each module has 3 sessions to be carried out in full. It is a systematic program, so the order of the sessions is regulated by the letters A, B and C for each module. The modules to be worked on correspond to the "low-level or languising" factors identified after the application of the positive mental health questionnaire (PMHQ). After the application of the PMHQ, people are grouped with the same module to work.
  Arms: Participants integrate the Mentis Plus+ program

SUMMARY:
The aim of this study is to evaluate the efficacy of a positive mental health program for adults, designated Mentis Plus+, in community. Our hypotheses are:

1. compared with the wait-list control group, the persons who join the experimental group and participate in the Mentis Plus+, will have more positive mental health on the end of the program;
2. in the Mentis Plus+ participants, positive mental health will be increased at the end of the program and at follow-up (three- six months later) and their psychological vulnerability will reduce.

ELIGIBILITY:
Inclusion Criteria:

* to be a participant aged ≥ 18;
* participant without a diagnosis of psychiatric pathology;
* agree to participate in the program by signing informed consent;
* participant with the "low-level or languising" in at least one factor of the positive mental health questionnaire

Exclusion Criteria:

* non-Portuguese speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive Mental Health Questionnaire (PMHQ) - moment 1 | PMHQ will be applied in the baseline of the Mentis Plus+ Program, to both groups
  The PMHQ consists of 39 items. In the PMHQ, values between 39 (minimum value) and 156 (maximum value) can be obtained, and higher the value obtained, lower the positive Mental Health level is. Therefore, we can categorize different levels of Positive Mental Health: High level or Flourishing (Results between 39-78), Intermediate level (Results between 79-117) and Low level or Languising (Results between 118-156).
Positive Mental Health Questionnaire (PMHQ) - moment 2 | PMHQ will be applied up to 18 weeks of the Mentis Plus + Program,to both groups
  The PMHQ consists of 39 items. In the PMHQ, values between 39 (minimum value) and 156 (maximum value) can be obtained, and higher the value obtained, lower the positive Mental Health level is. Therefore, we can categorize different levels of Positive Mental Health: High level or Flourishing (Results between 39-78), Intermediate level (Results between 79-117) and Low level or Languising (Results between 118-156).
Positive Mental Health Questionnaire (PMHQ) - moment 3 | The PMHQ will be reapplied for follow-up of the evaluation, after completion of the study, on average 3 months, in both groups
  The PMHQ consists of 39 items. In the PMHQ, values between 39 (minimum value) and 156 (maximum value) can be obtained, and higher the value obtained, lower the positive Mental Health level is. Therefore, we can categorize different levels of Positive Mental Health: High level or Flourishing (Results between 39-78), Intermediate level (Results between 79-117) and Low level or Languising (Results between 118-156).
Psychological Vulnerability Scale (PVS) - moment 1 | PVS will be applied in the baseline of the Mentis Plus+ Program, to both groups
  The PVS is a six-item scale. Each item is measured in a scale Frequency Likert five points (1-5), where a higher number corresponds to greater frequency (does not describe me at all = 1 to describes me very well = 5). Possible total scores range from 6 to 30, with higher scores indicating greater psychological vulnerability.
  greater psychological vulnerability.
Psychological Vulnerability Scale (PVS) - moment 2 | PVS will be applied up to 18 weeks of the Mentis Plus + Program,to both groups
  The PVS is a six-item scale. Each item is measured in a scale Frequency Likert five points (1-5), where a higher number corresponds to greater frequency (does not describe me at all = 1 to describes me very well = 5). Possible total scores range from 6 to 30, with higher scores indicating greater psychological vulnerability.
  greater psychological vulnerability.
Psychological Vulnerability Scale (PVS) - moment 3 | PVS will be reapplied for follow-up of the evaluation, after completion of the study, on average 3 months, in both groups
  The PVS is a six-item scale. Each item is measured in a scale Frequency Likert five points (1-5), where a higher number corresponds to greater frequency (does not describe me at all = 1 to describes me very well = 5). Possible total scores range from 6 to 30, with higher scores indicating greater psychological vulnerability.
  greater psychological vulnerability.

SECONDARY OUTCOMES:
Sociodemografic and clinical data - moment 1 | Sociodemografic and clinical data will be applied in the baseline of the Mentis Plus+ Program, to both groups
  Gender, age, marital status, educational level, professional bond, displacement of usual residence, years of professional practice, hours of work per week, history of mental illness, health behaviors in the last month, consumption of psychoactive substances
Sociodemografic and clinical data - moment 2 | Sociodemografic and clinical data will be applied up to 18 weeks of the Mentis Plus + Program,to both groups
  Gender, age, marital status, educational level, professional bond, displacement of usual residence, years of professional practice, hours of work per week, history of mental illness, health behaviors in the last month, consumption of psychoactive substances
Sociodemografic and clinical data - moment 3 | Sociodemografic and clinical data will be reapplied for follow-up of the evaluation, after completion of the study, on average 3 months, in both groups
  Gender, age, marital status, educational level, professional bond, displacement of usual residence, years of professional practice, hours of work per week, history of mental illness, health behaviors in the last month, consumption of psychoactive substances

CONTACTS AND LOCATIONS:
Locations (1):
- ACES Cavado I, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teixeira SMA, Ferre-Grau C, da Cruz Sequeira CA, Santos JM, Guerra MM, Lluch MT. Randomized Controlled Trial to Evaluate the Efficacy of Positive Mental Health Program for Adults: Study Protocol. Public Health Nurs. 2025 Jan-Feb;42(1):154-160. doi: 10.1111/phn.13427. Epub 2024 Oct 3. PMID 39359154